CLINICAL TRIAL: NCT04836871
Title: Clinical Research of Double Filtration Plasmapheresis Combined With Chemotherapy to Remove M Protein in Multiple Myeloma
Brief Title: Double Filtration Plasmapheresis Combined With Chemotherapy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fuling Zhou (Other)
Responsible Party: Sponsor-Investigator, Fuling Zhou, Head, Division of Hematology; Professor of Hematology; Doctoral advisor, Zhongnan Hospital
Organization: Zhongnan Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01
Record Dates: First submitted 2021-03-07; First posted 2021-04-08 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Double filtration plasmapheresis (DFPP) combined with chemotherapy (Experimental)
  Interventions: Combination Product: DFPP combined with chemotherapy

INTERVENTIONS:
Combination Product: DFPP combined with chemotherapy — Double filtration plasmapheresis combined with chemotherapy

SUMMARY:
Evaluation of double filtration plasmapheresis combined with chemotherapy for the treatment of abnormalities of M protein or renal function due to the multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Multiple myeloma patients who are diagnosed by bone marrow morphology and immunology
* Patients with stable condition after conventional treatment
* Patients with renal insufficiency or abnormal M protein
* Patients over 18 years of age
* Liver function: blood bilirubin ≤ 35μmol/L, enzymes aspartate transaminase (AST)/aka alanine aminotransferase (ALT) is less than 2 times the upper limit of normal
* Normal heart function
* Physical condition score 0-2 level (ECOG score)
* Obtain an informed consent form signed by the patient or family member

Exclusion Criteria:

* Allergies or obvious contraindications to any of the drugs involved in the plan
* Severe heart disease, including myocardial infarction and cardiac insufficiency.
* Suffering from other organ malignancies
* Active tuberculosis patients and HIV-positive patients
* At the same time suffering from other blood system diseases
* Pregnant or lactating women
* Able to understand or follow the research plan
* Past history of intolerance or allergy to similar drugs
* Patients under 18 years of age
* Participating in other clinical researchers at the same time
* There are any other circumstances that hinder the progress of the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-05-15 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
M protein clearance rate | 1hour
  before each treatment of Double filtration plasmapheresis (DFPP)
M protein clearance rate | 1hour
  after each treatment of DFPP
creatinine clearance rate | 1hour
  before each treatment of DFPP
creatinine clearance rate | 1hour
  after each treatment of DFPP
albumin concentration | 1hour
  before each treatment of DFPP
albumin concentration | 1hour
  after each treatment of DFPP
serum-free light chain levels | 1hour
  before each treatment of DFPP
serum-free light chain levels | 1hour
  after each treatment of DFPP
blood urea nitrogen | 1hour
  before each treatment of DFPP
blood urea nitrogen | 1hour
  after each treatment of DFPP
Platelet concentrations | 1hour
  before each treatment of DFPP
Platelet concentrations | 1hour
  after each treatment of DFPP

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes